CLINICAL TRIAL: NCT04347369
Title: a Retrospective Study of Neural Network Model to Dynamically Quantificate the Severity in COVID-19 Disease
Status: Completed | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy Director,Head of Oncology department, Principal Investigator, Clinical Professor, Xinqiao Hospital of Chongqing
Other Study IDs: XQonc-015
Record Dates: First submitted 2020-03-18; First posted 2020-04-15 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed group: The patients who were detected COVID-19 disease by RT-PCR and CT imaging.
  Interventions: Other: other

INTERVENTIONS:
Other: other — clinical diagnosis

SUMMARY:
The research aim to collect large samples of COVID-19 disease patients with clinical symptoms, laboratory and imaging examination data. Screening the biological indicators which are related to the occurrence of severe diseases. Then, investigators using artificial intelligence (AI) technology deep learning method to find a prediction model that can dynamically quantify COVID-19 disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients of COVID-19 disease confirmed by virus nucleic acid RT-PCR and CT

Exclusion Criteria:

* unconfirmed suspected cases
* Patients during pregnancy and lactation
* incomplete clinical data
* inestigators considered patients ineligible for the trial

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of COVID-19 disease
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
discrimination | up to 3 months
  The performance of our prediction model is evaluated with the receiver operating characteristic (ROC) curves, areas under the curves (AUCs) and concordance index (c-index).
Calibration | up to 3 months
  The calibration curves analysis is used to show error between the predicted clinical phenotype with prediction model and actual clinical phenotype.
Net benefit | up to 3 months
  Decision curve analysis was used to determine whether the models could be considered useful tools for clinical decisionmaking by comparing the net benefits at any threshold.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China